CLINICAL TRIAL: NCT04582526
Title: A Brief Body-mind-spirit Intervention to Promote Positive Emotions - a Pilot Trial
Brief Title: A Brief Body-mind-spirit Intervention to Promote Positive Emotions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Caritas Medical Centre, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UW 20-668
Record Dates: First submitted 2020-09-29; First posted 2020-10-09 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Emotions; Stress
Keywords: Personal well-being; Family well-being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): BMS program
  Interventions: Behavioral: BMS program

INTERVENTIONS:
Behavioral: BMS program — A BMS program with three components: relaxation exercises, healthy eating, expressive arts therapy

SUMMARY:
Integrating ICT in health promotion has been suggested to offer many advantages compared to traditional approaches to promote well-being. Research has shown the positive effects of a body-mind-spirit (BMS) approach in enhancing health and well-being. We will develop and assess a pilot trial involving a holistic BMS approach to promote positive emotion change, emotion regulation and self-awareness through an ICT-supported program in a community setting.

DETAILED DESCRIPTION:
The body-mind-spirit (BMS) approach views the three components as a connected, balanced system that interacts with one another harmoniously. With the well-established academic-community partnership between HKU and Caritas-Hong Kong, our pilot trial aims to build upon the previous experiences by Caritas-Hong Kong and investigate the feasibility and effectiveness of a BMS approach in enhancing positive emotions and well-being among community participants. This trial is an innovative attempt at conducting an ICT-supported online intervention with community participants. It would also help meet the urgent need for brief, community-based preventive mental health promotion, especially in the context of the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Chinese-speaking;
* Individuals aged 18 years and above;
* No history of diagnosed mental illness;
* Access to an internet-connected computer.

Exclusion Criteria:

* Individuals who cannot meet the inclusion criteria.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Positive emotion | Baseline and one month
  Change assessed by the Subjective Happiness Scale (SHS). The minimum and maximum of SHS are 4 to 24, respectively. A higher score means a better outcome.

SECONDARY OUTCOMES:
Stress level | Baseline and one month
  Change assessed by the Perceived Stress Scale (PSS). The minimum and maximum of SHS are 0 to 16, respectively. A higher score means a worse outcome.
Personal well-being | Baseline and one month
  Change assessed by a one-item Personal Happiness scale. The minimum and maximum of SHS are 0 to 10, respectively. A higher score means a better outcome.
Family well-being | Baseline and one month
  Change assessed by a 3-item Family well-being scale. The minimum and maximum are 0 to 30, respectively. A higher score means a better outcome.
Negative emotion | Baseline and one month
  Change assessed by the Patient Health Questionnaire-4. The minimum and maximum of SHS are 0 to 28, respectively. A higher score means a worse outcome.
Sleep quality | Baseline and one month
  Change assessed by the Insomnia Severity Index (ISI). The minimum and maximum of SHS are 0 to 28, respectively. A higher score means a worse outcome.
Knowledge and attitudes towards and practice of the holistic BMS health care approach | Baseline and one month
  Change assessed by outcome-based questions. A score of each question ranges from 1-5. A higher score a better outcome.
Perceived benefits of the BMS program | One month
  Assessed by outcome-based questions with categorical choices
Sharing of BMS with others | One month
  Assessed by outcome-based questions with categorical choices

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Y Lai, PhD, Principal Investigator — School of Nursing, The University of Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The minimal anonymized dataset will be available upon request to interested researchers. For interested researchers, please contact, Ms Shirley Sit (email shirlsit@hku.hk), (School of Public Health, The University of Hong Kong) for further information.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the study finished and the related papers were published
Access Criteria: The access should be requested through the written application with the reason of data used, and subject to the permission of principal investigator

REFERENCES:
- [Background] Chan C, Ho PS, Chow E. A body-mind-spirit model in health: an Eastern approach. Soc Work Health Care. 2001;34(3-4):261-82. doi: 10.1300/j010v34n03_02. PMID 12243428
- [Background] Ho RT, Sing CY, Wong VP. Addressing holistic health and work empowerment through a body-mind-spirit intervention program among helping professionals in continuous education: A pilot study. Soc Work Health Care. 2016 Nov-Dec;55(10):779-793. doi: 10.1080/00981389.2016.1231153. Epub 2016 Sep 22. PMID 27805500
- [Background] Lau BHP, Chow AYM, Ng TK, Fung YL, Lam TC, So TH, Chan JSM, Chan CHY, Zhou J, Tam MYJ, Tsang MW, Cheng NSY, Lim PFM, Chow SF, Chan CLW, Wong DFK. Comparing the efficacy of integrative body-mind-spirit intervention with cognitive behavioral therapy in patient-caregiver parallel groups for lung cancer patients using a randomized controlled trial. J Psychosoc Oncol. 2020 Jul-Aug;38(4):389-405. doi: 10.1080/07347332.2020.1722981. Epub 2020 Mar 9. PMID 32146876